CLINICAL TRIAL: NCT00508911
Title: An Open-label, Repeat-dose, Single-sequence Study to Investigate the Effects of Once-daily Repeat Oral Administration of GW876008 125mg on the Pharmacokinetics of the Combined Oral Contraceptive in Female Volunteers
Brief Title: A Study To Evaluate The Effect Of GW876008 On The Pharmacokinetics Of Oral Contraceptive Pills
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRH103002
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Social Phobia
Keywords: open-label,; oral contraceptive,; Combine Oral Contraceptives,; single-sequence,; volunteers; GW876008,; repeat-dose,; female,; pharmacokinetics,
MeSH Terms: conditions — Phobia, Social | interventions — GW 876008

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy female subjects (Experimental): Each subject will be administered a monophasic combined oral contraceptive (COC) containing ethinylestradiol 30 micrograms and levonorgestrel 150 micrograms for two complete cycles (Day 8 to Day 28) in Session 1. The subjects will be administered COC on Day 8 to Day 28 and GW876008 125 milligrams on Days 1 to 35 in Session 2.
  Interventions: Drug: GW876008; Drug: COC

INTERVENTIONS:
Drug: GW876008 — GW876008 tablets will be available as white to off-white coated tablets. Each subject will receive a single oral dose of GW876008, daily for up to 35 days in Session 2. GW876008 will be administered in the morning with a light breakfast.
  Other Names: GW876008 Oral Contraceptive
Drug: COC — COC containing ethinylestradiol 30 microgram and levonorgestrel 150 microgram will be administered in the morning with a light breakfast.

SUMMARY:
This study will be conducted in healthy female volunteers to investigate the effect of GW876008 on the pharmacokinetics of oral contraceptive pills.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential, who:

  * have been taking for at least 3 months a monophasic combined oral contraceptives (COC) (21 repeat-days administration + 7-days washout) containing ethinyloestradiol 30µg and levonorgestrel 150 µg;
  * are willing to continue a monophasic COC containing ethinyloestradiol 30µg and levonorgestrel 150 µg from at least the commencement of their last normal period prior to the first dose of study medication;
  * are willing to continue a monophasic COC containing ethinyloestradiol 30µg and levonorgestrel 150 µg until 14 days after last treatment or until the first normal period (defined as normal for the woman, both in terms of duration and quantity of menses) after last treatment, whichever is the longest.
* Women should have a regular menstrual cycle of approximately 4 weeks duration in the preceding 3 months.
* Females of childbearing potential will be required to use other adequate contraception, in addition to the COC
* Aged 18-45 years inclusive.
* Healthy subjects, defined as individuals who are free from clinically significant illness or disease as determined by their medical and psychiatric history (including family), physical examination, laboratory studies, and other tests.
* Body weight ≥ 45 kg for women and BMI within the range 18.5-29.9 kg/m2 inclusive;
* Demonstrates no evidence of active disease, physical or significant mental impairment.
* Self-administered Beck Depression Inventory II scale total score no greater than 9, and suicide question score of zero.
* Non-smoker (abstinence from smoking for at least 6 months before the start of the study).
* Agrees to abstain from ingesting caffeine or xanthine-containing products for 24 hours prior to the start of dosing until collection of the final pharmacokinetic sample.
* Agree to abstain from alcohol for 24 hours prior to the start of dosing until collection of the final pharmacokinetic sample.
* Normal electrocardiogram (subjects must have no clinically significant abnormalities on a 12-lead ECG and a 24 hour Holter ECG).
* Hormone assessments must be within normal range, at the pre-study assessment.
* Agree to remain in the clinic for the time defined in the protocol.
* Subject who has a history of peptic ulcer disease (PUD) with known aetiology must provide documentation by a gastroenterologist of the aetiology of the PUD and that effective treatment was provided with full eradication of ulcers and symptoms. For such subjects appropriate steps must also have been taken to minimize reoccurrence of risk (i.e. if PUD was nonsteroidal anti-inflammatory drug [NSAID] induced, the subject should no longer be taking NSAID medications; if cause was H. pylori, the subject should have been appropriately treated). Subjects with a history of PUD >10 years ago, without recurrence, may be included after discussion with the medical monitor even if documentation from treating physician is not available or aetiology unclear. See Section 6.3.6 for more details.
* Signed and dated written informed consent prior to admission to the study.
* The subject is able to understand and comply with protocol requirements,

Exclusion Criteria:

* As a result of any of the medical interview, physical examination or screening investigations the physician responsible considers the subject unfit for the study.
* Any clinical condition in which the COC is contra-indicated
* Female subjects who are currently or planning to become pregnant or lactating (from screening through at least 8 weeks after receiving study drug).
* The subject has a positive pre-study urine drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study HIV 1/2, Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Any history of suicidal attempts or behaviour.
* History of alcohol/drug abuse or dependence within 12 months of the study: history of regular alcohol consumption averaging > 14 drinks/week for women [1 drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits] within 6 months of screening.
* Consumption of grapefruit juice or grapefruit within 14 days prior to the first dose of study medication.
* Any history of an endocrine disorder including, but not limited to, diabetes or disorders of the hypothalamus, pituitary, adrenal, or thyroid glands, or gonadal disorder or dysfunction of the reproductive organs.
* Pepsinogen I, ACTH, cortisol, TSH, Total T4, Free T4 at screening/baseline outside > 5% of normal range.
* LFTs elevated above the reference range at pre-study screening that remain elevated with a repeat LFT
* Any other clinically significant laboratory abnormality.
* The subject has a screening ECG with values outside the ranges defined in the protocol
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 90 days or 5 half-lives, or twice the duration of the biological effect of any drug(whichever is longer) prior to the first dose of current study medication
* Other than prescribed COC, use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John'sWort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* History or presence of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* Where participation in study would result in donation of blood in excess of 500 mL within a 90 day period.
* Average daily caffeine intake equivalent to > 4 cups of coffee or > 6 cups of tea.
* A semi-supine systolic blood pressure less than 90mmHg or greater than 140mmHg or a semi-supine diastolic blood pressure of less than 50mmHg or greater than 90mmHg; or a radial pulse rate less than 40bpm or more than 90bpm.
* Subjects with positive faecal occult blood test.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2007-06-08 (Actual); Primary Completion 2007-10-22 (Actual); Study Completion 2007-10-22 (Actual)

PRIMARY OUTCOMES:
Blood level of oral contraceptive pills | measured over 24hrs on Day 28 of Period 1 and 2

SECONDARY OUTCOMES:
1)PK parameters of oral contraceptives | Day 28
2)PK parameters of GW876008 | Days 28 and 35 (Period2)
3)Blood level of sex hormones 4) Frequency of breakthrough bleeding 5) adverse event,12-lead ECG and vital signs and laboratory tests | (throughout study)
Ethinylestradiol and levonorgestrel blood levels to determine pharmacokinetic parameter | Session 1: Day 28 at pre-dose (-30 mins), 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24 hours post-dose. Session 2: Day 28 at pre-dose (-30 mins), 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24 hours post-dose. Days 30-35
Serum concentrations of LH, FSH. | Pre-dose on Days 8, 12 and 19
Serum concentration of progesterone and estradiol | Pre-dose on Days 25 and 28

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

REFERENCES:
- See also: Results for study CRH103002 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/CRH103002?search=study&search_terms=CRH103002#rs